CLINICAL TRIAL: NCT03209063
Title: The Role of Prothrombin Gene and Methylenetetrahydrofolate Reductase(MTHFR) Gene Polymorphisms as Risk Factors for Recurrent Miscarriage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mahran, principal investigator, Assiut University
Other Study IDs: TROPGP
Record Dates: First submitted 2017-07-01; First posted 2017-07-06 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Recurrent Miscarriage
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: 195 Patients having history of two or more miscarriages.
  Interventions: Diagnostic Test: polymerase chain reaction
- Group II: 90 healthy controls less than 35 years with no history of miscarriage and at least one uncomplicated full-term pregnancy
  Interventions: Diagnostic Test: polymerase chain reaction

INTERVENTIONS:
Diagnostic Test: polymerase chain reaction — diagnostic test as Polymerase chain reaction for detection of Prothrombin gene and methylenetetrahydrofolate reductase gene polymorphisms
  Other Names: homocysteine assay

SUMMARY:
Recurrent miscarriage is a pregnancy loss before 20 weeks of gestation. The recurrent pregnancy loss(RPL) usually occurring in the first trimester of gestation and its rate is quite high (15-20% even in full reproductive period) . In 2012, the American Society for Reproductive Medicine Practice Committee issued a statement that defined recurrent pregnancy loss as a disease distinct from infertility defined by two or more failed consecutive pregnancies.approximately 40% of couples will have an etiology identified that could be associated with their loss.

DETAILED DESCRIPTION:
Recurrent miscarriage is a pregnancy loss before 20 weeks of gestation. The recurrent pregnancy loss usually occurring in the first trimester of gestation and its rate is quite high (15-20% even in full reproductive period) . In 2012, the American Society for Reproductive Medicine Practice Committee issued a statement that defined recurrent pregnancy loss as a disease distinct from infertility defined by two or more failed consecutive pregnancies.approximately 40% of couples will have an etiology identified that could be associated with their loss.Thrombophilia is the tendency to develop thromboses due to inherited defects in the coagulation system.Thrombophilia was identified as a major cause of RPL,Because pregnancy is a hypercoagulable state, thromboembolism is the leading cause of antepartum and postpartum maternal mortality .The four most common genetic markers for thrombophilia are; prothrombin gene mutation(FII, G20210A), methylene tetra hydrofolate reductase mutations (MTHFR ,C677T and A1298C), factor V Leiden (FVL, G1691A) , and plasminogen activator inhibitor 1 (PAI-1) . Prothrombin G20210A refers to a human gene mutation that increases the risk of blood clots . Approximately 1 in 50 people in the white population in the United States and Europe has prothrombin thrombophilia. Study was conducted to evaluate the frequency of PT20210 among healthy Egyptians, (1.06%) had PT20210 G-A mutation.The variant causes elevated plasma prothrombin levels (hyperprothrombinemia), Prothrombin is the precursor to thrombin, which plays a key role in causing blood to clot (blood coagulation).Prothrombin G20210A can thus contribute to a state of hypercoagulability . Methylene tetra hydrofolate reductase (MTHFR) is the rate-limiting enzyme in the methyl cycle, and it is encoded by the Methylene tetra hydrofolate reductase gene. It was thought that deficient Methylene tetra hydrofolate reductase, by causing elevated homocysteine levels, led to an increased risk of venous thrombosis, coronary heart disease, and recurrent pregnancy loss . Previous studies suggested that percentage of PT20210 in patients with unexplained RPL is ( 10.9%),however searching literatures didn't find any estimation of this percentage in Egyptian population.

ELIGIBILITY:
Inclusion Criteria

1. Age less than 35 years.
2. History of two or more spontaneous miscarriages

Exclusion Criteria:

1. Age more than 35 years.
2. . Women with elevated level of TSH above (2.5 mIU/ml) and uncontrolled DM.
3. Women with autoimmune disorder (antiphospholipid antibody syndrome)with LA1/LA2 ratio more than( 1.2).
4. Women receiving oral contraceptive pills and anticoagulant drugs.

Ages: 17 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be conducted at Clinical Pathology Department,Women's Health Hospital ,Assiut University Hospital, Faculty of Medicine, Assiut University
Sampling Method: Non-Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The study will compare the percentage of prothrombin gene and MTHFR gene polymorphisms in cases with recurrent miscarriage and healthy control group. | 2 days
  using polymerase chain reaction Polymerase chain reaction

CONTACTS AND LOCATIONS:
Overall Officials: Ghada M Mahran, MD, Principal Investigator — Assiut University, Faculty of medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farahmand K, Totonchi M, Hashemi M, Reyhani Sabet F, Kalantari H, Gourabi H, Mohseni Meybodi A. Thrombophilic genes alterations as risk factor for recurrent pregnancy loss. J Matern Fetal Neonatal Med. 2016;29(8):1269-73. doi: 10.3109/14767058.2015.1044431. Epub 2015 Jul 2. PMID 26135458
- [Derived] Ahmed Abd Elhameed Z, Shaaban OM, Abd Elazeem HG, Abouelfadle A, Farghaly T, Mahran G, Seddik MI. Role of Prothrombin and Methylenetetrahydrofolate Reductase Gene Polymorphisms as well as Thrombophilia Markers, as Risk Factors for Unexplained Recurrent Miscarriage: A Case-Control Study. Int J Fertil Steril. 2025 Jan 5;19(1):36-43. doi: 10.22074/ijfs.2023.1986225.1418. PMID 39827389